CLINICAL TRIAL: NCT00820092
Title: A Phase 1,Dose Escalation Study to Compare the Safety, Tolerability,Pharmacokinetic and Pharmacodynamic Profiles of the 24-hour Intravenous Administration of Xerecept in Healthy Japanese and Caucasian Adult Volunteers
Brief Title: Xerecept Intravenous Dose Escalation in Japanese and Caucasian Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celtic Pharma Development Services (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Xerecept: CPDS 0805
Record Dates: First submitted 2008-12-14; First posted 2009-01-09 (Estimated); Last update posted 2013-07-30 (Estimated); Status verified 2013-07

CONDITIONS: Edema
Keywords: Xerecept; Pharmacokinetics; Japanese versus Caucasians
MeSH Terms: conditions — Edema

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Xerecept 1.0 (Active Comparator): 1.0 ug/kg/hr hCRF -24 hour IV infusion
  Interventions: Drug: Xerecept 1.0
- Xerecept 2.0 (Active Comparator): 2.0 ug/kg/hr-24 hour IV infusion
  Interventions: Drug: Xerecept 2.0
- Xerecept 3.0 (Active Comparator): 3.0 ug/kg/hr-24 hour infusion
  Interventions: Drug: Xerecept 3.0

INTERVENTIONS:
Drug: Xerecept 1.0 — 24 hour infusion
  Other Names: hCRF infusion; 1.0 ug/kg/hr
  Arms: Xerecept 1.0
Drug: Xerecept 2.0 — 24 hour infusion
  Other Names: hCRF infusion; 2.0 ug/kg/hr
  Arms: Xerecept 2.0
Drug: Xerecept 3.0 — 24 hour infusion
  Other Names: hCRF infusion; 3.0 ug/kg/hr
  Arms: Xerecept 3.0

SUMMARY:
1. To investigate the safety and tolerability of Xerecept during and following a 24-hour intravenous administration to healthy Japanese to healthy Japanese and Caucasian subjects
2. To compare the PK profile of hCRF during and following a 24-hour intravenous Xerecept administration between healthy Japanese and Caucasian subjects

DETAILED DESCRIPTION:
none needed

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female Japanese subjects who are citizens of Japan
* Healthy male and female Caucasian subjects
* Age range 20-45 years
* BMI >19 and <27 kg/m squared

Exclusion Criteria:

* Female subjects must not be pregnant at the time of study and use adequate birth control methods before,during and 4 weeks after the study
* Subjects must be negative for HCV and HIV
* Subjects must have negative urine tests for drugs of abuse and alcohol at screening
* Subjects must not have any clinically significant medical conditions

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2008-12; Primary Completion 2009-03 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Frequency and severity of AEs Clinical laboratory tests( chemistry,hematology,urinalysis) Physical exam and vital signs ECG AUC, Tmax Cmax Terminal half life AUC for cortisol concentration | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- West Coast Clinical Trials, Cypress, California, United States